CLINICAL TRIAL: NCT00579332
Title: Effects of Brassica or Indole-3-Carbinol on Prostatectomy Patients With PSA Recurrenc
Brief Title: Effects of Brassica or Indole-3-carbinol on Prostatectomy Patients With PSA Recurrence
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: American Institute of Cancer Prevention (Unknown)
Responsible Party: Principal Investigator, Jay Fowke, Associate Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 041001
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Biochemical Failure
Keywords: PSA; biochemical failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): one a day placebo
  Interventions: Dietary Supplement: brassica intervention
- 2 (Experimental): Brassica intake
  Interventions: Dietary Supplement: brassica intervention
- 3 (Experimental): indole-3-carbinol supplement
  Interventions: Dietary Supplement: brassica intervention

INTERVENTIONS:
Dietary Supplement: brassica intervention — diet and phyto-chemical intervention

SUMMARY:
Pilot and feasibility diet and phyto-agent intervention among healthy men at risk for prostate cancer progression.

ELIGIBILITY:
Inclusion Criteria:

* Men with PSA recurrence following prostatectomy

Exclusion Criteria:

* Not using exogenous hormones

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
change in blood PSA levels | 6 months

SECONDARY OUTCOMES:
monitor for health events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jay H Fowke, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt_University, Nashville, Tennessee, United States